CLINICAL TRIAL: NCT03047343
Title: Evolution of Two Cohorts of Children (Univentricular and Bi-ventricular Heart) After Strapping of the Pulmonary Artery
Status: Completed | Type: Observational
Sponsor: Pierre Wauthy (Other)
Responsible Party: Sponsor-Investigator, Pierre Wauthy, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-strapping
Record Dates: First submitted 2017-02-07; First posted 2017-02-08 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Congenital Heart Malformations
Keywords: pulmonary artery strapping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uni-ventricular reparation: All patients treated with pulmonary artery strapping between 2005 and 2016 at the Queen Fabiola Children Hospital. Patients benefiting from an uni-ventricular reparation.
  Interventions: Other: Retrospective data extraction in medical files
- Bi-ventricular reparation: All patients treated with pulmonary artery strapping between 2005 and 2016 at the Queen Fabiola Children Hospital. Patients benefiting from an bi-ventricular reparation.
  Interventions: Other: Retrospective data extraction in medical files

INTERVENTIONS:
Other: Retrospective data extraction in medical files — Retrospective data extraction in medical files

SUMMARY:
Pulmonary artery strapping is a surgical technique aimed at providing a palliative treatment to newborns suffering from congenital heart defects, characterized by an increase in blood flow and pulmonary blood pressure.

The intervention consists of placing a band around the pulmonary artery. This band causes an artificial stenosis, therefore inducing a reduction of the pulmonary arterial pressure. It acts as a first step, preparing the ground for a future definitive repair intervention.

It is mainly used in the context of septal defects, atrio-ventricular canal defects or uni-ventricular hearts.

The complications linked to strapping include, among others, the erosion of the band in the artery lumen, its migration and the obstruction of the pulmonary artery, a pulmonary valvular insufficiency, the obstruction of the coronary artery and an ineffective strapping.

The early mortality rate of pulmonary artery strapping after 1980 varies between 1.8% and 13.6%, while strapping readjustment rates oscillate around 20%. It is assumed that the mortality is linked to the nature of the cardial malformation (uni-ventricular or bi-ventricular) rather than the procedure itself.

This retrospective study aims to evaluate the intra-hospital and extra-hospital mortality rate of pulmonary artery strapping, as well as the readjustment rate within two groups of patients: those benefiting from an uni-ventricular cardiac reparation and those benefiting from a bi-ventricular cardiac reparation. The aim is to determine the short term mortality rate of the intervention and the incidence of complications within the hospital, within the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with pulmonary artery strapping between 2005 and 2016 at the Queen Fabiola Children Hospital

Exclusion Criteria:

* Outdated indications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with pulmonary artery strapping between 2005 and 2016 at the Queen Fabiola Children Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Date of birth | 12 years
  Date of birth of the patient
Sex | 12 years
  Sex of the patient
Weight | 12 years
  Weight of the patient at the time of the intervention
Exact diagnosis | 12 years
  Exact diagnosis at the time of the intervention
Exact date of intervention | 12 years
  Exact calender date of intervention
Total number of interventions | 12 years
  Total number of interventions
SpO2 | 12 years
  pre-surgery oxygen saturation
Date of death | 12 years
  If applicable, date of death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bellofatto Piazza, Principal Investigator — HUDERF; Pierre Wauthy, MD, Study Director — CHU Brugmann
Locations (1):
- HUDERF, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horowitz MD, Culpepper WS 3rd, Williams LC 3rd, Sundgaard-Riise K, Ochsner JL. Pulmonary artery banding: analysis of a 25-year experience. Ann Thorac Surg. 1989 Sep;48(3):444-50. doi: 10.1016/s0003-4975(10)62881-0. PMID 2476086
- [Background] Pinho P, Von Oppell UO, Brink J, Hewitson J. Pulmonary artery banding: adequacy and long-term outcome. Eur J Cardiothorac Surg. 1997 Jan;11(1):105-11. doi: 10.1016/s1010-7940(96)01049-4. PMID 9030797
- [Background] Valente AS, Mesquita F, Mejia JA, Maia IC, Maior MS, Branco KC, Pinto VC Jr, Carvalho W Jr. Pulmonary artery banding: a simple procedure? A critical analysis at a tertiary center. Rev Bras Cir Cardiovasc. 2009 Jul-Sep;24(3):327-33. doi: 10.1590/s0102-76382009000400011. English, Portuguese. PMID 20011878
- [Background] Takayama H, Sekiguchi A, Chikada M, Noma M, Ishizawa A, Takamoto S. Mortality of pulmonary artery banding in the current era: recent mortality of PA banding. Ann Thorac Surg. 2002 Oct;74(4):1219-23; discussion 1223-4. doi: 10.1016/s0003-4975(02)03900-0. PMID 12400772
- [Background] Yoshimura N, Yamaguchi M, Oka S, Yoshida M, Murakami H. Pulmonary artery banding still has an important role in the treatment of congenital heart disease. Ann Thorac Surg. 2005 Apr;79(4):1463; author reply 1463-4. doi: 10.1016/j.athoracsur.2003.12.113. No abstract available. PMID 15797113
- [Background] Brooks A, Geldenhuys A, Zuhlke L, Human P, Zilla P. Pulmonary artery banding: still a valuable option in developing countries? Eur J Cardiothorac Surg. 2012 Feb;41(2):272-6. doi: 10.1016/j.ejcts.2011.05.053. Epub 2011 Dec 12. PMID 21733709